CLINICAL TRIAL: NCT00974675
Title: A Double-Blind, Placebo Controlled Study to Assess the Pharmacokinetics, Safety and Tolerability of Multiple Intravenous Doses of 3 Dose Levels of CAT-354 in Subjects With Moderate Asthma
Brief Title: A Study to Assess Pharmacokinetics, Safety and Tolerability of Multiple Doses of CAT-354 in Subjects With Moderate Asthma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study recruitment was terminated before the planned number of subjects was enrolled in CAT-354 10 mg/kg group due to the slow recruitment rate.
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAT-354-0602; 2006-003199-36 (EudraCT Number)
Record Dates: First submitted 2009-09-08; First posted 2009-09-10 (Estimated); Results first posted 2017-05-02 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-03

CONDITIONS: Moderate Asthma
Keywords: Asthma; CAT-354; Tralokinumab
MeSH Terms: conditions — Asthma | interventions — tralokinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- CAT-354 1 mg/kg (Experimental): CAT-354 1 milligram/kilogram (mg/kg) of body weight intravenous infusion over 30 minutes on Day 0, 28 and 56.
  Interventions: Biological: CAT-354 1mg/kg
- CAT-354 5 mg/kg (Experimental): CAT-354 5 mg/kg of body weight intravenous infusion over 30 minutes on Day 0, 28 and 56.
  Interventions: Biological: CAT-354 5 mg/kg
- CAT-354 10mg/kg (Experimental): CAT-354 10 mg/kg of body weight intravenous infusion over 30 minutes on Day 0, 28 and 56.
  Interventions: Biological: CAT-354 10mg/kg
- Placebo (Placebo Comparator): Placebo matched to CAT-354 intravenous infusion over 30 minutes on Day 0, 28 and 56.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: CAT-354 1mg/kg — CAT-354 1 mg/kg of body weight intravenous infusion over 30 minutes on Day 0, 28 and 56.
  Other Names: Tralokinumab
  Arms: CAT-354 1 mg/kg
Biological: CAT-354 5 mg/kg — CAT-354 5 mg/kg of body weight intravenous infusion over 30 minutes on Day 0, 28 and 56.
  Other Names: Tralokinumab
  Arms: CAT-354 5 mg/kg
Biological: CAT-354 10mg/kg — CAT-354 10 mg/kg of body weight intravenous infusion over 30 minutes on Day 0, 28 and 56.
  Other Names: Tralokinumab
  Arms: CAT-354 10mg/kg
Other: Placebo — Placebo matched to CAT-354 intravenous infusion over 30 minutes on Day 0, 28 and 56.
  Arms: Placebo

SUMMARY:
The study includes participants with moderate asthma who were randomly assigned to receive the study medication (CAT-354) or placebo.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo controlled study. Following confirmation of eligibility, subjects with moderate asthma will be recruited sequentially to one of three dose groups and randomly assigned within dose group to either CAT-354 or placebo. Doses of the assigned treatment will be administered on three occasions 28 days apart. Follow up for pharmacokinetic blood sampling and safety will continue to Day 147 post-first dose (91 days post-third dose).

ELIGIBILITY:
Inclusion Criteria:

* Males or infertile females
* Subjects with asthma, well controlled on inhaled corticosteroid and taken as required (PRN) short acting beta 2 agonist therapy only
* Unchanged dose of inhaled corticosteroid for 3 months prior to Day 0 and no expected need for change in dose during study
* Forced expiratory volume in 1 second (FEV1) greater than or equal to 80% predicted at Screening (Baseline)
* 18-60 years
* General Practitioner diagnosis of asthma of 1 year's minimum duration (with respect to Day 0)
* No significant abnormality on clinical examination or medical history (excluding atopic skin signs, symptoms and history)
* 12-lead electrocardiogram with no clinical significant abnormality
* Clinical chemistry hematology and urinalysis results within the laboratory reference ranges or deemed not clinically significant by the Investigator
* A negative screen for drugs of abuse and alcohol
* Body weight between 50-120 kg
* Subjects aged between 18-40 years inclusive must have body mass index (BMI) 18-32 kilogram per square meter (kg/m^2) inclusive. Subjects aged between 41-60 years must have BMI between 18-30 kg/m^2 inclusive.

Exclusion Criteria:

* Active concomitant disease, with exception of eczema
* Expected onset of seasonal allergy before the administration of the last dose of study medication
* History of severe exacerbation within 3 years of Day 0
* Recorded use of inhaled short acting beta 2 agonist medication for symptoms within 14 days of Day 0 of: More than 6 doses per day on any 1 day or more than 3 doses per day on 6 or more days
* Any medication other than: inhaled short-acting beta 2 agonist, inhaled corticosteroids, topic eczema treatments (with the exception of fluorinated corticosteroid, dermatological preparations which are not permitted), hormone replacement therapy, vitamin preparation/food supplements, occasional use of proton pump inhibitors, ranitidine, cimetidine, antacids or over-the-counter analgesics
* Treatment within 6 months of Day 0 with any of the following: methylxanthines, inhaled cromones, leukotriene modifiers, anti- immunoglobulin E (IgE), anticholinergics, ketotifen, oral short acting B2 agonists, long-acting B2 agonists, oral or injected corticosteroids
* Treatment of atopic symptoms, other than eczema, within 4 weeks of Day 0
* History of medication that might carry-over effects into the study
* Previously received monoclonal antibody, or a similar related protein, that might sensitize to CAT-354
* Participation in another study within three months of the start of the study or 5 half lives of the previously administered investigational medicinal product (IMP), whichever is longer
* Lower respiratory tract infection within 4 weeks of Day-14
* Any acute illness in the two weeks before Day 0
* Current smokers, those who have smoked in previous year, and those with smoking history of greater than or equal to 10 pack years
* Considered by the investigator to be at risk of transmitting, through blood, the agents responsible for infectious diseases
* Blood donation (550 ml) in the previous 2 months
* Excessive intake of alcohol (more than 21 units a week for females or 28 units a week for males)
* The subject's general practitioner has suggested a reason the subject should not participate in the study
* The Investigator considers the subject should not take part for any reason.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2006-09-29 (Actual); Primary Completion 2007-08-03 (Actual); Study Completion 2007-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune LLC, Study Director — MedImmune LLC
Locations (1):
- Chiltern International Limited, Slough, Berkshire, United Kingdom

REFERENCES:
- [Background] Singh D, Kane B, Molfino NA, Faggioni R, Roskos L, Woodcock A. A phase 1 study evaluating the pharmacokinetics, safety and tolerability of repeat dosing with a human IL-13 antibody (CAT-354) in subjects with asthma. BMC Pulm Med. 2010 Jan 8;10:3. doi: 10.1186/1471-2466-10-3. PMID 20064211

RESULTS

PARTICIPANT FLOW:
Groups:
- CAT-354 10 mg/kg: CAT-354 10 mg/kg of body weight intravenous infusion over 30 minutes on Day 0, 28 and 56.
Period: Overall Study
Arm/Group | CAT-354 1 mg/kg | CAT-354 5 mg/kg | CAT-354 10 mg/kg | Placebo
Started | 8 | 8 | 3 | 4
Completed | 6 | 7 | 1 | 2
Not Completed | 2 | 1 | 2 | 2
Not completed — Adverse Event | 2 | 1 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Participant on holiday; unable to attend | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of investigational medicinal product (IMP: CAT-354 or placebo) including those who did not complete the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | CAT-354 1 mg/kg | CAT-354 5 mg/kg | CAT-354 10 mg/kg | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 3 | 4 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.4 (9.07) | 34.6 (7.58) | 43.3 (14.47) | 40.0 (13.04) | 38.3 (9.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 0 | 1
  Male | 8 | 8 | 2 | 4 | 22

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Serum Concentration (Cmax) for CAT-354 After First Dose
Time Frame: Pre-dose, 10 minutes and 12 hours post-end of infusion on Day 0; Day 4, 7, 14 and 21
Population: Pharmacokinetic (PK) population included all participants in the safety population for whom sufficient post-dose blood samples were taken to estimate a Cmax.
Measure: Mean (Standard Deviation); unit: microgram/milliliter (mcg/mL)
Arm/Group | CAT-354 1 mg/kg | CAT-354 5 mg/kg | CAT-354 10 mg/kg
Number analyzed (Participants) | 8 | 8 | 3
microgram/milliliter (mcg/mL) | 30.3 (5.18) | 156.8 (34.55) | 306.3 (31.39)

2. Primary Outcome: Maximum Observed Serum Concentration (Cmax) for CAT-354 After Second Dose
Time Frame: Pre-dose, 10 minutes and 12 hours post-end of infusion on Day 28; Day 35
Population: PK population included all participants in the safety population for whom sufficient post-dose blood samples were taken to estimate a Cmax. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | CAT-354 1 mg/kg | CAT-354 5 mg/kg | CAT-354 10 mg/kg
Number analyzed (Participants) | 7 | 7 | 1
mcg/mL | 35.0 (6.81) | 161.0 (32.81) | 298.0 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group.

3. Primary Outcome: Maximum Observed Serum Concentration (Cmax) for CAT-354 After Third Dose
Time Frame: Pre-dose, 10 minutes and 12 hours post-end of infusion on Day 56; Day 63, 84, 105 and 147
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | CAT-354 1 mg/kg | CAT-354 5 mg/kg | CAT-354 10 mg/kg
Number analyzed (Participants) | 6 | 7 | 1
mcg/mL | 41.1 (4.77) | 178.7 (25.41) | 393.0 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group.

4. Primary Outcome: Area Under the Serum Concentration Time Curve From Time Zero to Last Measurable Concentration (AUC[0 - t]) for CAT-354 After First Dose
Time Frame: Pre-dose, 10 minutes and 12 hours post-end of infusion on Day 0; Day 4, 7, 14 and 21
Population: PK population included all participants in the safety population for whom sufficient post-dose blood samples were taken to estimate a Cmax.
Measure: Mean (Standard Deviation); unit: (mcg*day)/mL
Arm/Group | CAT-354 1 mg/kg | CAT-354 5 mg/kg | CAT-354 10 mg/kg
Number analyzed (Participants) | 8 | 8 | 3
(mcg*day)/mL | 299.6 (42.03) | 1691.3 (302.70) | 3106.3 (719.25)

5. Primary Outcome: Area Under the Serum Concentration-Time Curve From Time Zero to Infinity (AUC[0 - Infinity]) for CAT-354 After First Dose
Description: AUC (0 - infinity) = Area under the serum concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - infinity). It is obtained from AUC (0 - t) plus AUC (t - infinity).
Time Frame: Pre-dose, 10 minutes and 12 hours post-end of infusion on Day 0; Day 4, 7, 14 and 21
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: (mcg*day)/mL
Arm/Group | CAT-354 1 mg/kg | CAT-354 5 mg/kg | CAT-354 10 mg/kg
Number analyzed (Participants) | 8 | 8 | 3
(mcg*day)/mL | 428.0 (83.33) | 2314.3 (392.91) | 3861.3 (662.42)

6. Primary Outcome: Apparent Terminal Elimination Phase Half-Life (t[1/2]el) for CAT-354 After First Dose
Description: Terminal elimination phase half-life is the time measured for the serum concentration to decrease by one half.
Time Frame: Pre-dose, 10 minutes and 12 hours post-end of infusion on Day 0; Day 4, 7, 14 and 21
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CAT-354 1 mg/kg | CAT-354 5 mg/kg | CAT-354 10 mg/kg
Number analyzed (Participants) | 8 | 8 | 3
days | 16.6 (2.67) | 16.1 (3.60) | 11.8 (1.86)

7. Primary Outcome: Clearance (CL) for CAT-354 After First Dose
Description: Clearance of a drug was a measure of the rate at which a drug was metabolized or eliminated by normal biological processes. Clearance was normalized by the body weight of the participant.
Time Frame: Pre-dose, 10 minutes and 12 hours post-end of infusion on Day 0; Day 4, 7, 14 and 21
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: (mL/day)/kilogram
Arm/Group | CAT-354 1 mg/kg | CAT-354 5 mg/kg | CAT-354 10 mg/kg
Number analyzed (Participants) | 8 | 8 | 3
(mL/day)/kilogram | 2.41 (0.45) | 2.23 (0.46) | 2.64 (0.42)

8. Primary Outcome: Volume of Distribution (Vd) for CAT-354 After First Dose
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. Volume of distribution was normalized to the body weight of the participant.
Time Frame: Pre-dose, 10 minutes and 12 hours post-end of infusion on Day 0; Day 4, 7, 14 and 21
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | CAT-354 1 mg/kg | CAT-354 5 mg/kg | CAT-354 10 mg/kg
Number analyzed (Participants) | 8 | 8 | 3
mL/kg | 56.7 (8.04) | 51.0 (10.36) | 44.0 (0.79)

9. Primary Outcome: Observed Serum Drug Concentration for CAT-354 28 Days (C28) After First Dose
Time Frame: Pre-dose on Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | CAT-354 1 mg/kg | CAT-354 5 mg/kg | CAT-354 10 mg/kg
Number analyzed (Participants) | 8 | 7 | 1
mcg/mL | 5.3 (1.33) | 27.1 (4.91) | 40.7 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group.

10. Primary Outcome: Observed Serum Drug Concentration for CAT-354 28 Days (C28) After Second Dose
Time Frame: Pre-dose on Day 56
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | CAT-354 1 mg/kg | CAT-354 5 mg/kg | CAT-354 10 mg/kg
Number analyzed (Participants) | 6 | 7 | 1
mcg/mL | 7.7 (1.63) | 36.0 (11.51) | 59.4 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group.

11. Primary Outcome: Observed Serum Concentration for CAT-354 28 Days (C28) After Third Dose
Time Frame: Day 84
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | CAT-354 1 mg/kg | CAT-354 5 mg/kg | CAT-354 10 mg/kg
Number analyzed (Participants) | 6 | 7 | 1
mcg/mL | 8.6 (1.99) | 40.6 (12.26) | 79.6 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group.

12. Secondary Outcome: Number of Participants Reporting Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to Day 147 that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Day 0 to Day 147
Population: Safety population included all participants who received at least 1 dose of IMP (CAT-354 or placebo) including those who did not complete the study.
Measure: Number; unit: participants
Groups:
- Placebp: Placebo matched to CAT-354 intravenous infusion over 30 minutes on Day 0, 28 and 56.
Arm/Group | CAT-354 1 mg/kg | CAT-354 5 mg/kg | CAT-354 10 mg/kg | Placebp
Number analyzed (Participants) | 8 | 8 | 3 | 4
participants
  TEAEs | 8 | 8 | 3 | 4
  TESAEs | 0 | 1 | 0 | 0

13. Primary Outcome: Accumulation Ratio (R0) for CAT-354
Description: Accumulation ratio is calculated as: R0 = AUC(56 - 84)/AUC(0 - 28) where AUC(0 - 28) and AUC(56 - 84) are the area under the serum concentration time curve over a dosage interval determined after the first dose (Day 0 to Day 28) and after the third dose (Day 56 to Day 84), respectively.
Time Frame: Pre-dose, 10 minutes and 12 hours post-end of infusion on Day 0 and 56; Pre-dose on Day 28; Day 4, 7, 14, 21, 63 and 84
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | CAT-354 1 mg/kg | CAT-354 5 mg/kg | CAT-354 10 mg/kg
Number analyzed (Participants) | 6 | 7 | 1
ratio | 1.58 (0.21) | 1.39 (0.10) | 1.67 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group.

ADVERSE EVENTS:
Time Frame: Day 0 to 147
Groups:
- 1 mg/kg: CAT-354 1 milligram/kilogram (mg/kg) of body weight intravenous infusion over 30 minutes on Day 0, 28 and 56.
- 5 mg/kg: CAT-354 5 mg/kg of body weight intravenous infusion over 30 minutes on Day 0, 28 and 56.
- 10 mg/kg: CAT-354 10 mg/kg of body weight intravenous infusion over 30 minutes on Day 0, 28 and 56.
Arm/Group | 1 mg/kg | 5 mg/kg | 10 mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/8 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 mg/kg (N=8) | 5 mg/kg (N=8) | 10 mg/kg (N=3) | Placebo (N=4)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 mg/kg (N=8) | 5 mg/kg (N=8) | 10 mg/kg (N=3) | Placebo (N=4)
Blepharospasm (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Feeling hot and cold (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Nasopharyngitis (Infections and infestations) | 5 (6) | 7 (10) | 2 (2) | 3 (4)
Pertussis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine analysis abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 4 (6) | 1 (1) | 2 (4)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Recruitment to the study was terminated before the planned number of participants was enrolled in CAT-354 10 mg/kg group due to the slow recruitment rate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.